CLINICAL TRIAL: NCT07366671
Title: SAvvywire for Pacing and Procedural Hemodynamics In Transcatheter Aortic Valve Replacement Evaluation; a Prospective Registry (SAPPHIRE)
Brief Title: SAvvywire for Pacing and Procedural Hemodynamics In Transcatheter Aortic Valve Replacement Evaluation
Acronym: SAPPHIRE
Status: Not yet recruiting | Type: Observational
Sponsor: dr Pim A.L. Tonino (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Sponsor-Investigator, dr Pim A.L. Tonino, Prof. Pim A.L. Tonino, MD, PhD, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Other Study IDs: SAPPHIRE - nWMO-2025.152; Funder (Other Grant/Funding Number: Haemonetics)
Record Dates: First submitted 2025-12-11; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation); Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (2):
- SavvyWire: TAVI procedures in which the SavvyWire is used as LV-guidewire.
- Other LV-guidwire: TAVI procedures in which another LV-guidewire (i.e. Confida or Safari) is used.

SUMMARY:
The goal of this observational study is to document which LV-guidewires are used during a TAVI (Transcatheter Aortic Valve Implantation) procedure and how their different functions perform.

A TAVI procedure is a minimally invasive treatment for aortic stenosis, where a new heart valve is inserted through a blood vessel in the groin. During this procedure, a wire (specifically, an LV-guidewire) is used to place the new heart valve. For this purpose, a regular LV-guidewire or a newer LV-guidewire with extra features, the Savvywire, can be used. All of these wires work well, are safe, and are already used in daily medical practice. Researchers will compare these LV-guidewires to see if the Savvywire adds additional value.

Patients aged 50 or older who undergo a TAVI procedure via the femoral artery (blood vessel in the groin) can participate. Participants will receive the usual care and standard follow-up, only their data will be collected and analyzed.

DETAILED DESCRIPTION:
Patients are asked for consent after the TAVI procedure. Procedural data is therefore collected retrospectively, while standard follow-up data (3 months after the procedure) is collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Accepted for transfemoral TAVI procedure by Heart team and TAVI team
* Transfemoral TAVI procedure with balloon-expandable or self-expandable TAVI platform
* Ability to understand and the willingness to provide written informed consent
* Patients scheduled for valve-in-valve procedures can be included
* Patients with bicuspid anatomy can be included

Exclusion Criteria:

* Patients planned for a non-transfemoral TAVI procedure
* Extremely horizontal aorta (aortic root angle >70 degrees)
* Extreme tortuosity at the level of the iliofemoral arteries, abdominal and/or thoracic aorta
* Inability to provide informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for participation in this registry are aged ≥50 years old presenting with symptomatic severe aortic valve stenosis and accepted for transfemoral TAVI procedure after consultation in the Heart team and TAVI team. A pre-procedural CT scan for TAVI sizing is required as standard of care. Both balloon-expandable and self-expandable TAVI platforms are allowed. Valve-in-valve procedures and procedures in bicuspid aortic valve anatomy can be included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Register which TAVI LV-guidewires are used in contemporary practice | At enrollment
  Register which type of TAVI LV-guidewire is used during the TAVI procedure (SavvyWire, Safari, Confida etc).
To register LV-aortic pressure gradients (mmHg) during each procedural step in the SavvyWire group. | Collected during TAVI procedure, extracted at enrollment
  With the SavvyWire, continuous hemodynamic pressure measurements can be performed during the procedure in the aorta and the left ventricle. Pressure measurements (mmHg) during the following procedural steps will be collected: baseline, pacing during predilatation, after predilatation, pacing during TAVI deployment, after TAVI deployment, after equilibration and drift check, after possibele postdilatation.
To correlate hemodynamic pressure gradient after each procedural step (predilatation, 80% TAVI deployment, postdilatation) to standard baseline CT assessment of valvular calcifications | At enrollment
Performance of the SavvyWire as LV-guidewire for TAVI device placement | At enrollment + after 3 months of standard follow-up
  Based on: guidewire kink yes/no, procedural success, complications during and after TAVI procedure and after standard 3 months follow-up (vascular complication, coronary obstruction, conversion to sternotomy, pacemaker, cva, mortality)
Performance of the SavvyWire in hemodynamic guidance | At enrollment
  Based on: succesfull hemodynamic registrations, drift check (delta between aortic pressure measurement of Savvywire and standard pigtail in aorta used during TAVI procedure), more postdilatation in Savvywire group compared to regular LV guidewire group.
Pacing performance of the SavvyWire | At enrollment
  Based on: pacing frequency, loss-of-capture, the need for RV pacing
To investigate the potential streamlining effect of the SavvyWire on TAVI workflow | At enrollment
  Based on: skin-to-skin time, total contrast volume (mL), amount of radiation exposure (total DAP, total Air Kerma)